CLINICAL TRIAL: NCT00235508
Title: The Efficacy of Eszopiclone 3 mg as Adjunctive Therapy in Subjects With Insomnia Related to Generalized Anxiety Disorder.
Brief Title: Safety and Efficacy of Eszopiclone in Patients With Generalized Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 190-902
Record Dates: First submitted 2005-10-06; First posted 2005-10-10 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Insomnia; Generalized Anxiety Disorder
Keywords: Insomnia; Anxiety; Generalized Anxiety Disorder
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Generalized Anxiety Disorder; Anxiety Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Escitalopram oxalate 10 mg at bedtime
  Interventions: Drug: Eszopiclone (Lunesta)
- 2 (Active Comparator): Eszopiclone 3 mg at bedtime
  Interventions: Drug: Eszopiclone (Lunesta)

INTERVENTIONS:
Drug: Eszopiclone (Lunesta) — Escitalopram oxalate 10 mg at bedtime; Eszopiclone 3 mg at bedtime
  Other Names: Lunesta

SUMMARY:
To determine the safety and efficacy of eszopiclone as adjunctive therapy in the treatment of insomnia in patients with insomnia related to Generalized Anxiety Disorder. All subjects will receive an approved anxiolytic agent and will be randomized to nightly therapy with either eszopiclone or placebo.

DETAILED DESCRIPTION:
An 8-week, randomized, double-blind, placebo-controlled, parallel-group adjunctive therapy trial. The study consists of subjects with insomnia related to Generalized Anxiety Disorder who will be treated for 10 weeks with open-label escitalopram oxalate 10 mg/day at bedtime, and randomized to receive either eszopiclone 3 mg nightly or placebo nightly for 8 weeks. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
* Subjects, between the ages of 18 and 64 years inclusive
* Subjects with Generalized Anxiety Disorder (GAD)
* Subjects with insomnia related to GAD.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420 (Actual)
Dates: Start 2005-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The change from baseline in subjective sleep latency averaged over the double-blind treatment period. | 8 weeks

SECONDARY OUTCOMES:
Change from baseline in subjective total sleep time averaged over the double blind treatment period. | 8 weeks

CONTACTS AND LOCATIONS:
Locations (64):
- United States (64):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Irvine, California
  - La Mesa, California
  - National City, California
  - Oceanside, California
  - Orange, California
  - Pasadena, California
  - Redlands, California
  - Riverside, California
  - San Diego, California
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Coral Springs, Florida
  - Fort Lauderdale, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - St. Petersburg, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Smyrna, Georgia
  - Northfield, Illinois
  - Indianapolis, Indiana
  - Owensboro, Kentucky
  - Baltimore, Maryland
  - Rockville, Maryland
  - Braintree, Massachusetts
  - Brighton, Massachusetts
  - Brockton, Massachusetts
  - Cambridge, Massachusetts
  - Watertown, Massachusetts
  - St Louis, Missouri
  - Kenilworth, New Jersey
  - Piscataway, New Jersey
  - Brooklyn, New York
  - Lawrence, New York
  - New York, New York
  - Durham, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - Bismarck, North Dakota
  - Beachwood, Ohio
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Middleburg Heights, Ohio
  - Eugene, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Moon Township, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scotland, Pennsylvania
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Austin, Texas
  - Houston, Texas
  - Richardson, Texas
  - San Antonio, Texas
  - Wichita Falls, Texas
  - Falls Church, Virginia
  - Richmond, Virginia
  - Middleton, Wisconsin

REFERENCES:
- [Result] Fava M, Schaefer K, Huang H, Wilson A, Iosifescu DV, Mischoulon D, Wessel TC. A post hoc analysis of the effect of nightly administration of eszopiclone and a selective serotonin reuptake inhibitor in patients with insomnia and anxious depression. J Clin Psychiatry. 2011 Apr;72(4):473-9. doi: 10.4088/JCP.09m05131gry. Epub 2010 Nov 2. PMID 21208574
- [Derived] Pollack M, Kinrys G, Krystal A, McCall WV, Roth T, Schaefer K, Rubens R, Roach J, Huang H, Krishnan R. Eszopiclone coadministered with escitalopram in patients with insomnia and comorbid generalized anxiety disorder. Arch Gen Psychiatry. 2008 May;65(5):551-62. doi: 10.1001/archpsyc.65.5.551. PMID 18458207